CLINICAL TRIAL: NCT03291509
Title: Remote Delivery of Weight Management for Adults With Intellectual and Developmental Disabilities (IDD)
Brief Title: Remote Delivery of Weight Management for Adults With IDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00140653; R01DK114121-01 (NIH)
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: weight loss; weight management
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person Group (Active Comparator): Participants randomized to this group will have a health educator to their house for in-person meetings. Participants will use paper forms to track progress in other parts of the study. Participants will be asked follow the Enhanced Stop Light Diet (eSLD) and take part in structured physical activity each week.
  Interventions: Behavioral: In-person Meetings; Behavioral: Enhanced Stop Light Diet; Behavioral: Physical Activity
- Computer Group (Experimental): Participants randomized to this group will use an iPad to talk to the health educator via video conference meetings. Participants will use the iPad to track progress in other parts of the study. Participants will be asked follow the Enhanced Stop Light Diet (eSLD) and take part in structured physical activity each week.
  Interventions: Behavioral: Video Conference Meetings; Behavioral: Enhanced Stop Light Diet; Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Video Conference Meetings — Individual video conferencing with a health educator using an iPad.
  Arms: Computer Group
Behavioral: In-person Meetings — Individual face-to-face (FTF) meetings with a health educator.
  Arms: In-person Group
Behavioral: Enhanced Stop Light Diet — Diet composed of healthy, pre-packaged meals, balance of fruits, vegetables, and low calories snacks, and shakes. Participants and study partners will be trained to use a color coded chart which categorize foods based on the Stop Light system (green, yellow, red) to assist in meal planning, grocery shopping, decisions regarding snack foods, and compliance with the diet in special situations such as eating away from home (restaurants, parties, etc.).
  Other Names: eSLD
Behavioral: Physical Activity — Participants will be asked to complete a set amount of time of moderate-to-vigorous physical activity each week. Participants in the Computer group will be asked to attend remote exercise sessions 2 times a week.

SUMMARY:
The purpose of this study is to compare different weight loss programs in people with IDD to see which program works better.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate IDD as determined by a Community Service Provider operating in Kansas under the auspices of a Community Developmental Disability Organization (CDDO). Participants will be judged competent to provide informed consent by their CDDO, or will have a guardian with power of attorney.
* Ability to provide assent, regardless of guardian consent.
* BMI of 25 to 45 kg/m2
* Sufficient functional ability to understand directions, communicate preferences (e.g. foods), wants (e.g. more to eat/drink), and needs (e.g. assistance with food preparation) through spoken language
* Living at home with a parent/guardian, or in a supported living environment with a caregiver who assists with food shopping, meal planning, and meal preparation and agrees to serve as a study partner
* No plans to relocate outside the study area over the next 24 months
* Internet access in the home

Exclusion Criteria:

* Unable to participate in moderate-to-vigorous physical activity (MVPA)
* Insulin dependent diabetes
* Participation in a weight management program involving diet and physical activity in the past 6 months
* Serious food allergies, consuming special diets (vegetarian, Atkins etc.), aversion to common foods (e.g., unwilling to consume dairy products, vegetables), diagnosis of Prader-Willi Syndrome
* Pregnancy during the previous 6 months, currently lactating or planned pregnancy in the following 24 months.
* Serious medical risk, e.g., cancer, recent heart attack, stroke, angioplasty
* Unwilling to be randomized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2022-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, PhD, Principal Investigator — University of Kansas Medical Center; Lauren T Ptomey, PhD, RD, LD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Ptomey LT, Washburn RA, Sherman JR, Mayo MS, Krebill R, Szabo-Reed AN, Honas JJ, Helsel BC, Bodde A, Donnelly JE. Remote delivery of a weight management intervention for adults with intellectual disabilities: Results from a randomized non-inferiority trial. Disabil Health J. 2024 Apr;17(2):101587. doi: 10.1016/j.dhjo.2024.101587. Epub 2024 Jan 22. PMID 38272776
- [Derived] Ptomey LT, Washburn RA, Mayo MS, Greene JL, Lee RH, Szabo-Reed AN, Honas JJ, Sherman JR, Donnelly JE. Remote delivery of weight management for adults with intellectual and developmental disabilities: Rationale and design for a 24 month randomized trial. Contemp Clin Trials. 2018 Oct;73:16-26. doi: 10.1016/j.cct.2018.08.010. Epub 2018 Aug 24. PMID 30145269

RESULTS

PARTICIPANT FLOW:
Groups:
- Face to Face: Participants randomized to this group will have a health educator to their house for in-person meetings. Participants will use paper forms to track progress in other parts of the study. Participants will be asked follow the Enhanced Stop Light Diet (eSLD) and take part in structured physical activity each week.
  In-person Meetings: Individual face-to-face (FTF) meetings with a health educator.
  Enhanced Stop Light Diet: Diet composed of healthy, pre-packaged meals, balance of fruits, vegetables, and low calories snacks, and shakes. Participants and study partners will be trained to use a color coded chart which categorize foods based on the Stop Light system (green, yellow, red) to assist in meal planning, grocery shopping, decisions regarding snack foods, and compliance with the diet in special situations such as eating away from home (restaurants, parties, etc.).
  Physical Activity: Participants will be asked to complete a set amount of time of moderate-to-vigorous physical activity each week. Participants in the Computer group will be asked to attend remote exercise sessions 2 times a week.
- Remote Delivery: Participants randomized to this group will use an iPad to talk to the health educator via video conference meetings. Participants will use the iPad to track progress in other parts of the study. Participants will be asked follow the Enhanced Stop Light Diet (eSLD) and take part in structured physical activity each week.
  Video Conference Meetings: Individual video conferencing with a health educator using an iPad.
  Enhanced Stop Light Diet: Diet composed of healthy, pre-packaged meals, balance of fruits, vegetables, and low calories snacks, and shakes. Participants and study partners will be trained to use a color coded chart which categorize foods based on the Stop Light system (green, yellow, red) to assist in meal planning, grocery shopping, decisions regarding snack foods, and compliance with the diet in special situations such as eating away from home (restaurants, parties, etc.).
  Physical Activity: Participants will be asked to complete a set amount of time of moderate-to-vigorous physical activity each week. Participants in the Computer group will be asked to attend remote exercise sessions 2 times a week.
Period: Overall Study
Arm/Group | Face to Face | Remote Delivery
Started | 60 | 60
6 Months | 53 | 57
18 Months | 39 | 48
Completed | 33 | 46
Not Completed | 27 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Face to Face | Remote Delivery | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (11.7) | 30.6 (8.0) | 32.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 63
  Male | 25 | 32 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 55 | 56 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 49 | 54 | 103
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Weight (kg) [Mean (Standard Deviation); unit: kg] | 101.5 (27.5) | 94.4 (25.8) | 97.9 (26.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight (kg)
Description: Change in weight (kg) from baseline to 6 months
Time Frame: Change from Baseline to Month 6
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Face to Face | Remote Delivery
Number analyzed (Participants) | 53 | 57
kg | -2.1 (6.7) | -4.9 (7.8)

2. Secondary Outcome: Change in Weight (kg)
Description: Change in weight across the 24 month study
Time Frame: Change from Baseline to Month 24
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Face to Face | Remote Delivery
Number analyzed (Participants) | 33 | 46
kg | -2.3 (10.1) | -4.5 (10.3)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Face to Face | Remote Delivery
All-Cause Mortality (participants affected / at risk) | 1/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/60
Other Adverse Events (participants affected / at risk) | 3/60 | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Face to Face (N=60) | Remote Delivery (N=60)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Choking
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Face to Face (N=60) | Remote Delivery (N=60)
Broken Bone (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03291509/Prot_SAP_000.pdf